CLINICAL TRIAL: NCT04725318
Title: An Observational Study to Determine Feasibility and Validity of Esophageal and Transpulmonary Pressure Measurements During One Lung Ventilation
Brief Title: Esophageal Pressure Measurements During One-lung Ventilation
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Maximilian S Schaefer, Associate Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2020P-000811
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Surgery; One-lung Ventilation
Keywords: One-lung ventilation; Electrical Impedance Tomography; Thoracic Surgery; Esophageal manometry; Transpulmonary Pressure; Lung-protective ventilation
MeSH Terms: interventions — One-Lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: One-lung ventilation — One-lung ventilation as part of routine clinical care for patients undergoing thoracic surgery under general anesthesia

SUMMARY:
The investigators will assess the feasibility and validity of esophageal pressure measurements during one-lung ventilation in the lateral position for surgery by comparing to lung collapse estimated from electrical impedance tomography during a PEEP trial.

DETAILED DESCRIPTION:
In this prospective cohort study, the investigators will assess the feasibility of esophageal pressure measurements during general anesthesia with one-lung ventilation in patients undergoing non-cardiac intrathoracic surgery, which is typically conducted in the lateral position. The investigators will measure esophageal pressure with an esophageal balloon catheter. The investigators will compare esophageal pressure measurements to lung collapse estimated by Electrical Impedance Tomography (EIT).

Patients will be equipped with the EIT belt before induction of anesthesia, and a one-minute EIT recording during spontaneous breathing will be conducted. Anesthesia will be induced as to institutional standards and upon the discretion of the attending anesthesiologist. After placement of a double-lumen endotracheal tube, the esophageal balloon catheter will be placed.

* After placement of the esophageal catheter, esophageal pressure, transpulmonary pressure, airway pressure and flow and EIT signal will be recorded ("baseline").
* When the patient has been positioned for surgery (typically in the lateral position), a second recording of the above parameters is conducted ("lateral"). One-lung ventilation will then be initiated and a third measurement ("OLV") is made.
* During the third measurement, a decremental positive end-expiratory pressure trial will be conducted to correlate the measured esophageal pressure to the positive end-expiratory pressure where lung collapse is detected from EIT.
* Before surgery, the EIT belt is opened and removed from the surgical field to avoid interference.
* If feasible, when surgery is finished, before reversal of neuromuscular blockade and extubation, a final recording of EIT, esophageal pressure, transpulmonary pressure, airway pressure and flow will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing non-cardiac surgery with OLV

Exclusion Criteria:

* COPD
* Active respiratory infection
* Prior lung resection
* Prior esophageal/gastric surgery
* Esophageal varices
* Patients under effective anticoagulation at time of surgery
* Pacemaker/ICD
* Pregnancy
* Inability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing non-cardiac surgery requiring one-lung ventilation under general anesthesia as part of clinical routine
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Esophageal pressure at lung collapse | During one-lung ventilation
  Esophageal pressure during one-lung ventilation in the lateral position at beginning lung collapse as measured by electrical impedance tomography during a decremental PEEP titration

SECONDARY OUTCOMES:
Esophageal Pressure | During one-lung ventilation
  Esophageal Pressure during one-lung ventilation in the lateral position at airway closure as assessed by pressure-volume curves
Esophageal Pressure | During two-lung ventilation in the lateral position
  Esophageal Pressure during two-lung ventilation in the lateral position at airway closure as assessed by pressure-volume curves
Esophageal Pressure | During two-lung ventilation in the supine position
  Esophageal Pressure during two-lung ventilation in the supine position at airway closure as assessed by pressure-volume curves
Optimum PEEP | During one-lung ventilation
  PEEP during PEEP titration that provides optimum trade-off between lung collapse and overdistension, as measured by Electrical Impedance Tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No